CLINICAL TRIAL: NCT02445807
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Parallel Group Study of the Efficacy and Safety of DFD-06 Cream in the Treatment of Moderate to Severe Plaque Psoriasis for 14 Days
Brief Title: A Study of the Efficacy and Safety of DFD-06 Cream in the Treatment of Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD06-CD-005
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Chronic Stable Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD-06 cream (Experimental): DFD-06 Cream will be applied to subjects with moderate plaque psoriasis twice daily for 14 days.
  Interventions: Drug: DFD06-Cream
- Vehicle Cream (Placebo Comparator): Vehicle Cream will be applied to subjects with moderate plaque psoriasis twice daily for 14 days.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: DFD06-Cream — Twice daily topical application for 14 days.
  Other Names: Clobetasol propionate Cream, 0.025%
  Arms: DFD-06 cream
Drug: Vehicle Cream — Twice daily topical application for 14 days.
  Arms: Vehicle Cream

SUMMARY:
This study will compare the efficacy and safety of DFD-06 Cream to Vehicle Cream for topical treatment of moderate to severe plaque psoriasis after 3, 7, and 14 days of treatment.

DETAILED DESCRIPTION:
This study will be a multicenter (approximately 30 sites), randomized, vehicle-controlled, double-blind, and parallel group design. Approximately 264 subjects with moderate to severe plaque psoriasis will be randomized to treatment with DFD-06 Cream or Vehicle Cream. Subjects will use study product twice daily for 14 days. Subject visits are scheduled at Screening, Baseline (Day 1) and Days 4, 8, and 15. Clinical determinations of disease severity will be performed using the total sign score (TSS) for the target lesion and Investigator Global Assessment (IGA) for overall severity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands the study procedures and agrees to participate by giving written informed consent. Subjects must be willing to authorize use and disclosure of protected health information collected for the study.
2. Subject must be at least 18 years of age.
3. Subject must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.
4. Subject with psoriasis involving 3% or greater BSA, not including the face, scalp, groin, axillae and other intertriginous areas.
5. Subject must have an IGA grade of 3 or 4 (moderate to severe) at the Baseline Visit.
6. Female subjects of childbearing potential must agree to use contraception during the study which can include abstinence with an adequate secondary option should the subject become sexually active. All women of childbearing potential must complete a urine pregnancy test (test must have a sensitivity of at least 25mIU/ml for human chorionic gonadotropin) at the Baseline Visit (Visit 2) and the test result must be negative to be eligible for enrollment.
7. Subject must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
3. Presence of pigmentation, extensive scarring, or pigmented lesions or sunburn which could interfere with the rating of efficacy parameters.
4. History of psoriasis unresponsive to biological or topical treatments.
5. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
6. Use within 180 days prior to Baseline Visit of biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, secukinumab, or alefacept).
7. Have received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.
8. Use within 60 days prior to the Baseline Visit of: 1) systemic or topical immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) or 3) oral retinoids (e.g., acitretin, isotretinoin).
9. Use within 30 days prior to the Baseline Visit of: 1) systemic steroids, 2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy. Inhaled, intraocular, and intranasal steroids are allowed.
10. Use within 14 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene), 2) topical retinoids (e.g., tazarotene, tretinoin) or 3) topical corticosteroids.
11. Subjects who have participated in a study of an investigational drug 60 days prior to the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr Reddy's Laboratories Inc
Locations (30):
- United States (30):
  - Site 101, Birmingham, Alabama
  - Site 103, Mobile, Alabama
  - Site 130, Mesa, Arizona
  - Site 116, Phoenix, Arizona
  - Site 125, Tucson, Arizona
  - Site 120, North Hollywood, California
  - Site 114, San Diego, California
  - Site 127, Santa Monica, California
  - Site 128, Clearwater, Florida
  - Site 115, Miami, Florida
  - Site 118, Indianapolis, Indiana
  - Site 110, Louisville, Kentucky
  - Site 105, Glenn Dale, Maryland
  - Site 111, Warren, Michigan
  - Site 113, Fridley, Minnesota
  - Site 123, Saint Joseph, Missouri
  - Site 106, Newington, New Hampshire
  - Site 104, Albuquerque, New Mexico
  - Site 117, Stony Brook, New York
  - Site 124, High Point, North Carolina
  - Site 109, Winston-Salem, North Carolina
  - Site 129, Johnston, Rhode Island
  - Site 119, Anderson, South Carolina
  - Site 102, Greenville, South Carolina
  - Site 108, Austin, Texas
  - Site 122, Houston, Texas
  - Site 107, Plano, Texas
  - Site 112, Draper, Utah
  - Site 126, Spokane, Washington
  - Site 121, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DFD-06 Cream | Vehicle Cream
Started | 176 | 89
Completed | 176 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-06 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 176 | 89 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 70 | 222
  >=65 years | 24 | 19 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 38 | 103
  Male | 111 | 51 | 162
Region of Enrollment [Number; unit: participants]
  United States | 176 | 89 | 265

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Percentage of Subjects With Treatment Success)
Description: The primary efficacy endpoint is the percentage of subjects with treatment success (defined as IGA = 0 or 1 and at least a 2 grade reduction from Baseline) at the Day 15 visit.
  The primary analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: Day 15 Visit
Measure: Number; unit: percentage of participants
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 176 | 89
percentage of participants | 30.1 | 9.7

2. Secondary Outcome: The Percent Change in Body Surface Area of Psoriasis
Description: The percent change from baseline in Body Surface Area at Day 15. The analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: From Baseline to Day 15
Measure: Mean (Standard Deviation); unit: percentage change in body surface area
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 176 | 89
percentage change in body surface area | -25.1 (36.60) | -7.4 (20.28)

3. Secondary Outcome: The Percentage of Subjects With Treatment Success at the Day 8 Visit.
Description: The percentage of subjects with treatment success (defined as IGA = 0 or 1 and at least a 2 grade reduction from Baseline) at Day 8.
  The analysis was done with multiple imputations. Results are combined analyses from 5 imputed data sets.
Time Frame: At Day 8 Visit
Measure: Number; unit: percentage of participants
Arm/Group | DFD-06 Cream | Vehicle Cream
Number analyzed (Participants) | 176 | 89
percentage of participants | 14.2 | 1.6

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | DFD-06 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/176 | 0/89
Other Adverse Events (participants affected / at risk) | 27/176 | 26/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-06 Cream (N=176) | Vehicle Cream (N=89)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-06 Cream (N=176) | Vehicle Cream (N=89)
Heart Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
application site discolouration (General disorders) | 4 (4) | 0 (0)
Application Site Fissure (General disorders) | 1 (1) | 5 (5)
Application Site Pain (General disorders) | 12 (12) | 11 (11)
Application Site Pruritus (General disorders) | 5 (5) | 14 (14)
Application site Rash (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No